CLINICAL TRIAL: NCT05778682
Title: Decannulation of Tracheostomy Cannula Based on Suctioning Frequency and High-flow Oxygen Protocol in the Intensive Care Unit
Acronym: DECAP-ICU
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Université de Sherbrooke (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2022-4213
Record Dates: First submitted 2023-01-16; First posted 2023-03-21 (Actual); Last update posted 2023-03-21 (Actual); Status verified 2023-03

CONDITIONS: Tracheostomy Weaning

STUDY DESIGN:
Masking Description: None, patients and physicians will know the protocol
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Suction based protocol (Experimental): Weaning protocol based on suctioning frequency. Once the weaning of mechanical ventilation, the patients in this arm will be on high-flow nasal canula. The canula will be remove if the decannulation conditions are met (if the patient require less than 2 aspirations in 8 hours for 24 consecutive hours)
  Interventions: Procedure: Suctioning based protocol
- Usual care (Other): Usual care will mainly base on the capping trial.
  Interventions: Procedure: Usual Care

INTERVENTIONS:
Procedure: Suctioning based protocol — cf. arm The necessity of suctioning will be assed continuously by the nurses, respiratory therapist and the medical team. If the patient require 2 or less aspiration each 8 hours for 24 hours straight, an attempt of decanalution will be done.
  Arms: Suction based protocol
Procedure: Usual Care — Usual care in our center is tolerance to a capping trial.
  Arms: Usual care

SUMMARY:
In the DECAP-ICU trial, the investigators will be focusing on the impact of a new weaning tracheostomy technique based on suctioning frequency compared to the standard practice of capping tolerance.

ELIGIBILITY:
Inclusion Criteria:

* Weaning from mechanical ventilation for at least 24 hours
* Randomisation must be done in 24 hours of the mechanical ventilation weaning.

Exclusion Criteria:

* Sabadell > 2
* Contraindication of decannulation : Glasgow Coma Scale <6, severe dysphagia, non permeable respiratory tracks, neuromuscular disease (expect for the ICU weakness) and long term tracheostomy.

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2023-03-20 (Estimated); Primary Completion 2024-02-01 (Estimated); Study Completion 2025-02-01 (Estimated)

PRIMARY OUTCOMES:
Time to decannulation | Frome date of randomisation to the date of the actual decannulation or to the date of death, whichever comes first, assessed up to 48 months.
  Time between the randomisation and the decannulation

SECONDARY OUTCOMES:
Time to decannulation criteria | From date of randomisation to the date when the criteria of decannulation are met or to the date of death, whichever comes first, assessed up to 48 months.
  Time between the randomisation and the criteria of decannulation
Length of stay ICU | From admission to the date when the patient quit the ICU, through study completion, average of 6 to 12 months.
  Lenght of stay in the ICU.
Length of stay hospital | From admission to the date when the patient is discharge of the hospital, through study completion, average of 6 to 12 months.
  Length of stay in the hospital
ICU readmission | Through study completion, average of 6 to 12 months.
  ICU readmission
Decannulation failure | Through study completion, average of 6 to 12 months.
  Necessity of reimplantation of a tracheostomy after the decannulation
Mechanical Ventilation weaning failure | Through study completion, average of 6 to 12 months.
  Necessity of starting mechanical ventilation once the randomisation is started
Adverses effects | Through study completion, average of 6 to 12 months.
  Pneumonia, sepsis, septic shock
Mortality | Through study completion, average of 6 to 12 months.
  All cause mortality

CONTACTS AND LOCATIONS:
Locations (1):
- Université de Sherbrooke, Sherbrooke, Quebec, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Abe T, Madotto F, Pham T, Nagata I, Uchida M, Tamiya N, Kurahashi K, Bellani G, Laffey JG; LUNG-SAFE Investigators and the ESICM Trials Group. Epidemiology and patterns of tracheostomy practice in patients with acute respiratory distress syndrome in ICUs across 50 countries. Crit Care. 2018 Aug 17;22(1):195. doi: 10.1186/s13054-018-2126-6. PMID 30115127
- [Background] Hosokawa K, Nishimura M, Egi M, Vincent JL. Timing of tracheotomy in ICU patients: a systematic review of randomized controlled trials. Crit Care. 2015 Dec 4;19:424. doi: 10.1186/s13054-015-1138-8. PMID 26635016
- [Background] Mahmood K, Wahidi MM. The Changing Role for Tracheostomy in Patients Requiring Mechanical Ventilation. Clin Chest Med. 2016 Dec;37(4):741-751. doi: 10.1016/j.ccm.2016.07.013. Epub 2016 Oct 14. PMID 27842753
- [Background] Spataro E, Durakovic N, Kallogjeri D, Nussenbaum B. Complications and 30-day hospital readmission rates of patients undergoing tracheostomy: A prospective analysis. Laryngoscope. 2017 Dec;127(12):2746-2753. doi: 10.1002/lary.26668. Epub 2017 May 23. PMID 28543108
- [Background] Simon M, Metschke M, Braune SA, Puschel K, Kluge S. Death after percutaneous dilatational tracheostomy: a systematic review and analysis of risk factors. Crit Care. 2013 Oct 29;17(5):R258. doi: 10.1186/cc13085. PMID 24168826
- [Background] Mitchell RB, Hussey HM, Setzen G, Jacobs IN, Nussenbaum B, Dawson C, Brown CA 3rd, Brandt C, Deakins K, Hartnick C, Merati A. Clinical consensus statement: tracheostomy care. Otolaryngol Head Neck Surg. 2013 Jan;148(1):6-20. doi: 10.1177/0194599812460376. Epub 2012 Sep 18. PMID 22990518
- [Background] Ceriana P, Carlucci A, Navalesi P, Rampulla C, Delmastro M, Piaggi G, De Mattia E, Nava S. Weaning from tracheotomy in long-term mechanically ventilated patients: feasibility of a decisional flowchart and clinical outcome. Intensive Care Med. 2003 May;29(5):845-8. doi: 10.1007/s00134-003-1689-z. Epub 2003 Mar 13. PMID 12634987
- [Background] Natalini D, Grieco DL, Santantonio MT, Mincione L, Toni F, Anzellotti GM, Eleuteri D, Di Giannatale P, Antonelli M, Maggiore SM. Physiological effects of high-flow oxygen in tracheostomized patients. Ann Intensive Care. 2019 Oct 7;9(1):114. doi: 10.1186/s13613-019-0591-y. PMID 31591659
- [Background] Stripoli T, Spadaro S, Di Mussi R, Volta CA, Trerotoli P, De Carlo F, Iannuzziello R, Sechi F, Pierucci P, Staffieri F, Bruno F, Camporota L, Grasso S. High-flow oxygen therapy in tracheostomized patients at high risk of weaning failure. Ann Intensive Care. 2019 Jan 7;9(1):4. doi: 10.1186/s13613-019-0482-2. PMID 30617626
- [Background] Singer M, Deutschman CS, Seymour CW, Shankar-Hari M, Annane D, Bauer M, Bellomo R, Bernard GR, Chiche JD, Coopersmith CM, Hotchkiss RS, Levy MM, Marshall JC, Martin GS, Opal SM, Rubenfeld GD, van der Poll T, Vincent JL, Angus DC. The Third International Consensus Definitions for Sepsis and Septic Shock (Sepsis-3). JAMA. 2016 Feb 23;315(8):801-10. doi: 10.1001/jama.2016.0287. PMID 26903338
- [Background] Charlson ME, Pompei P, Ales KL, MacKenzie CR. A new method of classifying prognostic comorbidity in longitudinal studies: development and validation. J Chronic Dis. 1987;40(5):373-83. doi: 10.1016/0021-9681(87)90171-8. PMID 3558716
- [Background] Durbin CG Jr. Tracheostomy: why, when, and how? Respir Care. 2010 Aug;55(8):1056-68. PMID 20667153
- [Background] Trouillet JL, Collange O, Belafia F, Blot F, Capellier G, Cesareo E, Constantin JM, Demoule A, Diehl JL, Guinot PG, Jegoux F, L'Her E, Luyt CE, Mahjoub Y, Mayaux J, Quintard H, Ravat F, Vergez S, Amour J, Guillot M. Tracheotomy in the intensive care unit: guidelines from a French expert panel. Ann Intensive Care. 2018 Mar 15;8(1):37. doi: 10.1186/s13613-018-0381-y. PMID 29546588
- [Background] Yang A, Gray ML, McKee S, Kidwai SM, Doucette J, Sobotka S, Yao M, Iloreta A. Percutaneous versus surgical tracheostomy: timing, outcomes, and charges. Laryngoscope. 2018 Dec;128(12):2844-2851. doi: 10.1002/lary.27334. Epub 2018 Oct 3. PMID 30284256
- [Background] Adly A, Youssef TA, El-Begermy MM, Younis HM. Timing of tracheostomy in patients with prolonged endotracheal intubation: a systematic review. Eur Arch Otorhinolaryngol. 2018 Mar;275(3):679-690. doi: 10.1007/s00405-017-4838-7. Epub 2017 Dec 19. PMID 29255970
- [Background] Pandian V, Miller CR, Schiavi AJ, Yarmus L, Contractor A, Haut ER, Feller-Kopman DJ, Mirski MA, Morad AH, Carey JP, Hillel AT, Maragos CS, Bhatti NI. Utilization of a standardized tracheostomy capping and decannulation protocol to improve patient safety. Laryngoscope. 2014 Aug;124(8):1794-800. doi: 10.1002/lary.24625. Epub 2014 Apr 4. PMID 24473939
- [Background] Hernandez Martinez G, Rodriguez ML, Vaquero MC, Ortiz R, Masclans JR, Roca O, Colinas L, de Pablo R, Espinosa MD, Garcia-de-Acilu M, Climent C, Cuena-Boy R. High-Flow Oxygen with Capping or Suctioning for Tracheostomy Decannulation. N Engl J Med. 2020 Sep 10;383(11):1009-1017. doi: 10.1056/NEJMoa2010834. PMID 32905673
- [Background] Wan X, Wang W, Liu J, Tong T. Estimating the sample mean and standard deviation from the sample size, median, range and/or interquartile range. BMC Med Res Methodol. 2014 Dec 19;14:135. doi: 10.1186/1471-2288-14-135. PMID 25524443
- [Background] Fernandez R, Serrano JM, Umaran I, Abizanda R, Carrillo A, Lopez-Pueyo MJ, Rascado P, Balerdi B, Suberviola B, Hernandez G; Sabadell Score Study Group. Ward mortality after ICU discharge: a multicenter validation of the Sabadell score. Intensive Care Med. 2010 Jul;36(7):1196-201. doi: 10.1007/s00134-010-1825-5. Epub 2010 Mar 11. PMID 20221748
- [Background] Williams R, Rankin N, Smith T, Galler D, Seakins P. Relationship between the humidity and temperature of inspired gas and the function of the airway mucosa. Crit Care Med. 1996 Nov;24(11):1920-9. doi: 10.1097/00003246-199611000-00025. PMID 8917046
- [Background] Hasani A, Chapman TH, McCool D, Smith RE, Dilworth JP, Agnew JE. Domiciliary humidification improves lung mucociliary clearance in patients with bronchiectasis. Chron Respir Dis. 2008;5(2):81-6. doi: 10.1177/1479972307087190. PMID 18539721
- [Background] Parke R, McGuinness S, Eccleston M. Nasal high-flow therapy delivers low level positive airway pressure. Br J Anaesth. 2009 Dec;103(6):886-90. doi: 10.1093/bja/aep280. Epub 2009 Oct 20. PMID 19846404
- [Background] Groves N, Tobin A. High flow nasal oxygen generates positive airway pressure in adult volunteers. Aust Crit Care. 2007 Nov;20(4):126-31. doi: 10.1016/j.aucc.2007.08.001. Epub 2007 Oct 10. PMID 17931878
- [Background] Parke RL, McGuinness SP. Pressures delivered by nasal high flow oxygen during all phases of the respiratory cycle. Respir Care. 2013 Oct;58(10):1621-4. doi: 10.4187/respcare.02358. Epub 2013 Mar 19. PMID 23513246
- [Background] Parke RL, Eccleston ML, McGuinness SP. The effects of flow on airway pressure during nasal high-flow oxygen therapy. Respir Care. 2011 Aug;56(8):1151-5. doi: 10.4187/respcare.01106. Epub 2011 Apr 15. PMID 21496369
- [Background] Sim MA, Dean P, Kinsella J, Black R, Carter R, Hughes M. Performance of oxygen delivery devices when the breathing pattern of respiratory failure is simulated. Anaesthesia. 2008 Sep;63(9):938-40. doi: 10.1111/j.1365-2044.2008.05536.x. Epub 2008 Jun 6. PMID 18540928
- [Background] Ritchie JE, Williams AB, Gerard C, Hockey H. Evaluation of a humidified nasal high-flow oxygen system, using oxygraphy, capnography and measurement of upper airway pressures. Anaesth Intensive Care. 2011 Nov;39(6):1103-10. doi: 10.1177/0310057X1103900620. PMID 22165366